CLINICAL TRIAL: NCT02052609
Title: An Extension Study of KHK4827 in Subjects With Plaque Psoriasis (Psoriasis Vulgaris, Psoriatic Arthritis), Pustular Psoriasis (Generalized) and Psoriatic Erythroderma
Brief Title: A Phase 3 Clinical Study of KHK 4827
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4827-005
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2019-11

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis; Pustular; Psoriasis, Palmaris Et Plantaris; Psoriatic Erythroderma
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK4827 140mg SC (Experimental)
  Interventions: Drug: KHK4827 140mg SC
- KHK4827 210mg SC (Experimental)
  Interventions: Drug: KHK4827 210mg SC

INTERVENTIONS:
Drug: KHK4827 140mg SC — Experimental1:KHK4827 140mg subcutaneous injection
  Arms: KHK4827 140mg SC
Drug: KHK4827 210mg SC — Experimental2:KHK4827 210mg subcutaneous injection
  Arms: KHK4827 210mg SC

SUMMARY:
This study is designed to evaluate the safety and efficacy of long-term exposure to KHK4827 in subjects with plaque psoriasis (psoriasis vulgaris, psoriatic erythroderma) who have completed Study 4827-003 (Study 003)and in subjects with pustular psoriasis (generalized) or psoriatic erythroderma who have completed the Study 4827-004 (Study 004).

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed the written informed consent form to participate in this study
* Subject has completed the week 52 evaluation either in Study 003 or 004

Exclusion Criteria:

* Subject has had a serious infection, defined as requiring systemic treatment with antibiotics or antivirals (excluding oral administration)
* Subject has been judged to be ineligible for participation in the study by the investigators/sub investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01-28 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence and types of adverse events and adverse reactions | 28 weeks
Anti-KHK4827 antibody | 28 weeks

SECONDARY OUTCOMES:
Change in psoriasis area and severity index (PASI) compared to the data obtained before the first dose of investigational product in this study. | 28 weeks
Percent improvement in PASI | 28 Weeks
PASI 50, 75, 90, and 100 | 28 Weeks
Static physician's global assessment (sPGA) of "0 (clear) or 1(almost clear)" | 28 Weeks
sPGA of "0 (clear) | 28 weeks
Change in body surface area involvement (BSA) of lesion | 28 weeks
Clinical Global Impression (CGI) | 28 weeks
American College of Rheumatology (ACR) 20 | 28 weeks
Pustular symptom score | 28 weeks
Serum KHK4827 concentration | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Kirin, Chiyoda-ku, Tokyo, Japan